CLINICAL TRIAL: NCT01377753
Title: MR Image Guided Focal Therapy in Prostate Cancer
Brief Title: MR Image Guided Therapy in Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Peter Pinto, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 110158; 11-C-0158
Record Dates: First submitted 2011-06-18; First posted 2011-06-21 (Estimated); Results first posted 2022-02-01 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Prostate Cancer; Prostatic Neoplasms
Keywords: Toxicity; Thermal Ablation/Damage; Localized Prostate Cancer; Laser Ablation; PSA Levels; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Arm 1/Magnetic Resonance (MR) Thermal Image Guided Laser Ablation (Experimental): Eligible subjects will undergo MR thermal image guided laser ablation of all biopsy proven areas of prostate cancer using one or multiple laser probes during a single procedure lasting approximately two hours in duration.
  Interventions: Device: Visualase Thermal Therapy System

INTERVENTIONS:
Device: Visualase Thermal Therapy System — Used for performing Laser Induced Thermal Therapy to destroy malignant or unwanted tissue by delivering laser energy sufficient to cause coagulation and necrosis of the tissue.

SUMMARY:
Background:

- One way to treat prostate cancer is to use a laser to direct extreme heat to a small area of the prostate. The heat destroys tumor cells but does not affect healthy tissue. Doctors want to see if magnetic resonance imaging (MRI) can be used to improve this treatment. MRI will be used to help locate tumor cells and guide the laser during surgery. However, MRI-guided laser therapy has not been used to treat many people with prostate cancer. More studies are needed to see whether it can destroy tumor cells permanently.

Objectives:

- To test the safety and effectiveness of treating prostate tumors with laser therapy guided by magnetic resonance imaging.

Eligibility:

- Men at least 18 years of age who have prostate cancer that can be seen with an MRI and has not spread to other parts of the body.

Design:

* Participants will be screened with a physical exam and medical history. They will also have blood tests and imaging studies, and will complete questionnaires about their health.
* Participants will have the MRI-guided laser treatment in the hospital. The doctor will use the MRI to control how much energy is delivered by the laser and how much tissue is destroyed. The entire procedure usually takes from 1.5 to 3 hours.
* After the treatment, participants will have a catheter put in to keep the bladder emptied. The catheter will stay in for 1 to 7 days. Drugs to prevent infection and bladder spasms will be given. Participants will leave the hospital once they are well enough to go home.
* Participants will have follow-up visits 3, 6, 9, 12, 18, 24, and 36 months after the therapy. They will have physical exams, and blood and urine tests. They will also answer questionnaires. Participants will have MRI scans 6, 12, 24, and 36 months after the therapy. They will have a prostate biopsy to see if there is any tumor every 12 months for the first 2 years. Another biopsy may be done in the third year.

DETAILED DESCRIPTION:
Background:

* Pilot study is designed to evaluate the safety and feasibility of thermal laser ablation of focal prostate tumors.
* Prostate cancer is relatively slow growing, with doubling times for local tumors estimated at 2 to 4 years.
* Some prostate cancers prove to be small, low grade, and noninvasive and they appear to pose little risk to the life or health of the host. Recent patient series suggest that 20% to 30% of men undergoing radical prostatectomy have pathologic features in the radical prostatectomy specimen consistent with an insignificant or indolent cancer which poses little threat to life or health.
* We propose that patients with low volume and low grade disease can be best served with focal ablation of the visible prostate cancer without the side effects of urinary incontinence and erectile dysfunction associated with radiation therapy or radical surgery.

Objectives:

Primary Objective:

-To determine feasibility and safety of magnetic resonance image-guided focal laser ablation of biopsy confirmed and magnetic resonance (MR) visible prostate cancer.

Eligibility:

* Greater than 18 years of age
* Organ confined prostate cancer, observed on MR, and confirmed by Transrectal biopsy
* Preoperative workup as dictated by the National Comprehensive Cancer Network (NCCN).org prostate cancer guidelines
* Prostate-specific antigen (PSA) < 15 ng or PSA density < 0.15 ng/ml in patients with a PSA > 15 ng

Design:

* Pilot study, testing feasibility, safety and tolerability of thermal ablation of focal prostate cancer
* It is anticipated that 15 patients will be accrued for this study

ELIGIBILITY:
* INCLUSION CRITERIA:
* Men greater than 18 years of age
* Organ confined clinical T1C or clinical T2a prostate cancer that is visualized on magnetic resonance (MR) imaging
* Prostate cancer is diagnosed by transrectal ultrasound guided standard 12 core biopsy or MR image guided biopsies

  * Gleason Score less than or equal to 7 (3+4), less than or equal to 3 cores positive in a standard 12 core biopsy or less than or equal to 4 cores positive on MR image guided biopsy where in 2 cores are taken from each of the two magnetic resonance imaging (MRI) target lesions
  * If the standard biopsy cores are positive, they must be from the same location in the prostate as MR Lesion was biopsied and proven to be cancer. (Left / Right, Base, Mid Gland, Apex).
* MRI obtained within 6 months of ablation
* Metastatic Disease work up as per National Comprehensive Cancer Network (NCCN) guidelines (www.nccn.org). Bone scan indicated to r/o metastatic disease if [clinical T1 and prostate-specific antigen (PSA) > 20 or T2 and PSA > 10]
* PSA less than or equal to 15 ng/ml or PSA density less than or equal to 0.15 ng/ml(2) in patients with a PSA > 15 ng/ml
* The patient has given written informed consent after the nature of the study and alternative treatment options have been explained.
* Patients who present with local recurrence or residual tumor after prostate cancer treatment which is visible on MRI.

EXCLUSION CRITERIA:

* The presence of 3 or more MR Visible lesions positive on biopsy
* The presence of extra capsular, seminal vesical invasion or metastatic disease.
* Patient is unable to tolerate MRI (foreign body, i.e. pacemaker or other implanted device; claustrophobia; inability to tolerate rectal coil; etc.)
* Patient with inability to follow up
* Acute urinary tract infection
* Lower urinary tract symptoms defined by a International Prostate symptom score (IPSS) >20
* Patients with renal insufficiency with an estimated glomerular filtration (EGF) <= 30 are excluded, due to they will not be able to undergo gadolinium enhance MRI.
* Patients with Uncontrolled Coagulopathies who are at increased risk of bleeding.
* Altered mental status preventing consent or answering questions during conduct of the trial will be excluded for safety purposes.
* Other serious illnesses according to the Principal Investigator (PI): involving the cardiac, respiratory, central nervous system (CNS), renal or hepatic organ systems, which would preclude study completion or impede the determination of causality of any complications experienced during the conduct of this study.
* A Standard 12 core biopsy positive for cancer with no corresponding MR targeted lesion positive for cancer in the same general region of the prostate (Right Apex, Right Mid Gland, Right Base, Left Base, Left Mid Gland, Left Apex)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2011-08-12 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2018-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter A Pinto, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andriole GL, Crawford ED, Grubb RL 3rd, Buys SS, Chia D, Church TR, Fouad MN, Gelmann EP, Kvale PA, Reding DJ, Weissfeld JL, Yokochi LA, O'Brien B, Clapp JD, Rathmell JM, Riley TL, Hayes RB, Kramer BS, Izmirlian G, Miller AB, Pinsky PF, Prorok PC, Gohagan JK, Berg CD; PLCO Project Team. Mortality results from a randomized prostate-cancer screening trial. N Engl J Med. 2009 Mar 26;360(13):1310-9. doi: 10.1056/NEJMoa0810696. Epub 2009 Mar 18. PMID 19297565
- [Background] Adolfsson J. Watchful waiting and active surveillance: the current position. BJU Int. 2008 Jul;102(1):10-4. doi: 10.1111/j.1464-410X.2008.07585.x. Epub 2008 Apr 14. No abstract available. PMID 18422774
- [Result] Schroder FH, Hugosson J, Roobol MJ, Tammela TL, Ciatto S, Nelen V, Kwiatkowski M, Lujan M, Lilja H, Zappa M, Denis LJ, Recker F, Berenguer A, Maattanen L, Bangma CH, Aus G, Villers A, Rebillard X, van der Kwast T, Blijenberg BG, Moss SM, de Koning HJ, Auvinen A; ERSPC Investigators. Screening and prostate-cancer mortality in a randomized European study. N Engl J Med. 2009 Mar 26;360(13):1320-8. doi: 10.1056/NEJMoa0810084. Epub 2009 Mar 18. PMID 19297566
- [Result] Mehralivand S, George AK, Hoang AN, Rais-Bahrami S, Rastinehad AR, Lebastchi AH, Ahdoot M, Siddiqui MM, Bloom J, Sidana A, Merino MJ, Choyke PL, Shih JH, Turkbey B, Wood BJ, Pinto PA. MRI-guided focal laser ablation of prostate cancer: a prospective single-arm, single-center trial with 3 years of follow-up. Diagn Interv Radiol. 2021 May;27(3):394-400. doi: 10.5152/dir.2021.20095. PMID 34003127
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2011-C-0158.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1/Magnetic Resonance (MR) Thermal Image Guided Laser Ablation
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Arm 1/Magnetic Resonance (MR) Thermal Image Guided Laser Ablation
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.86 (7.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15
Median Prostate-Specific Antigen (PSA) [Median (Full Range); unit: ng/mL] | 6.19 [2.16 to 14.5]
Median Baseine Tumor Volume [Median (Full Range); unit: cm(3)] | 0.55 [0.19 to 3.27]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One Grade 1 Adverse Event, More Than One Grade 1 Adverse Event, and One Grade 2 Adverse Event
Description: Adverse events were assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). Grade 1 is mild and Grade 2 is moderate.
Time Frame: For all participants enrolled over the time frame of the study including follow up time is approximately 65 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1/Magnetic Resonance (MR) Thermal Image Guided Laser Ablation
Number analyzed (Participants) | 15
Participants
  One Grade 1 Adverse Event | 4
  More Than One Grade 1 Adverse Event | 2
  One Grade 2 Adverse Event | 4

2. Secondary Outcome: Mean Change in Prostate Specific Antigen (PSA) From Baseline Prior to Salvage Treatment or at the Conclusion of the Study Time Frame if There Was No Salvage Treatment
Description: A single difference was calculated between the PSA value measured at baseline and either (1) the PSA value measured just prior to a salvage treatment or (2) the PSA value measured at the conclusion of the study time frame (if no salvage treatment was necessary).
Time Frame: From date participant is enrolled to completion of post-ablation monitoring, approximately 3 years.
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Arm 1/Magnetic Resonance (MR) Thermal Image Guided Laser Ablation
Number analyzed (Participants) | 15
ng/mL | -2.5 (0.6)

3. Secondary Outcome: Mean Change in Prostate Specific Antigen Density (PSAD) From Baseline During Study Time Frame
Description: A single difference was calculated between the PSA density at baseline and either (1) the PSA density just prior to a salvage treatment or (2) the PSA density at the conclusion of the study time frame (if no salvage treatment was necessary).
Time Frame: From date participant is enrolled to completion of post-ablation monitoring, approximately 3 years.
Measure: Mean (Standard Deviation); unit: ng/dL/mL
Arm/Group | Arm 1/Magnetic Resonance (MR) Thermal Image Guided Laser Ablation
Number analyzed (Participants) | 15
ng/dL/mL | 0.114 (0.07)

4. Secondary Outcome: Mean Change in Quality of Life (QoL) From Baseline Prior to Salvage Treatment or at the Conclusion of the Study Time Frame if There Was No Salvage Treatment
Description: The outcome of laser ablation for treatment of prostate cancer for each participant was assessed by Quality of Life (QoL) questionnaire at clinic appointments. Specifically, patients are asked "How would you feel if you had to live with your urinary condition the way it is now, no better, no worse, for the rest of your life?" A score is then provided on a scale of 0 (delighted) to 5 (unhappy). The change in QoL from baseline was determined by calculating the difference between the baseline score and either the score just prior to a salvage treatment or the last measurement obtained at the conclusion of the study time frame.
Time Frame: From date participant is enrolled to completion of post-ablation monitoring, approximately 3 years.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Arm 1/Magnetic Resonance (MR) Thermal Image Guided Laser Ablation
Number analyzed (Participants) | 15
score on a scale | 0 (0.2)

5. Secondary Outcome: Mean Change in International Prostate Symptom Score (IPSS) From Baseline Over Follow-Up Visits Prior to Salvage Treatment or Across All Follow-up Visits During Study Time Frame if There Was No Salvage Treatment
Description: The outcome of laser ablation for treatment of prostate cancer for each participant was assessed by International Prostate Symptom Score (IPSS) questionnaire at clinic appointments. Specifically, patients are asked about seven domains of lower urinary tract symptoms (incomplete emptying, frequency, intermittency, urgency, weak stream, straining, and nocturia) and provide scores for each domain from 0 (not at all) to 5 (almost always) to describe how often they experience each symptom. Therefore, each domain is scored from 0 to 5. The scores are then totaled (summed). Therefore, the total score could range from 0 to 35. For both individual domain scores and the total score, a higher score indicates more severe symptoms. The change in IPSS from baseline was determined by calculating the difference between the baseline score and either the score just prior to a salvage treatment or the last measurement obtained at the conclusion of the study time frame.
Time Frame: From date participant is enrolled to completion of post-ablation monitoring, approximately 3 years.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Arm 1/Magnetic Resonance (MR) Thermal Image Guided Laser Ablation
Number analyzed (Participants) | 15
score on a scale | -1 (0.9)

6. Secondary Outcome: Mean Change in Sexual Health Inventory for Men (SHIM) From Baseline Over Follow-Up Visits Prior to Salvage Treatment or Across All Follow-up Visits During Study Time Frame if There Was No Salvage Treatment
Description: The outcome of laser ablation for treatment of prostate cancer for each participant was assessed by Sexual Health Inventory for Men (SHIM) questionnaire at clinic appointments. Specifically, patients are asked six questions about sexual health and erectile function and provide scores for each question from 0 (not at all) to 5 (almost always) to describe how often they experience each symptom. Therefore, each question is scored from 0 to 5. The scores are then totaled (summed). Therefore, the total score could range from 0 to 30. For both individual question scores and the total score a lower score indicates more severe symptoms. The mean change in SHIM from baseline was determined by calculating the difference between the baseline score and either the score just prior to a salvage treatment or the last measurement obtained at the conclusion of the study time frame.
Time Frame: From date participant is enrolled to completion of post-ablation monitoring, approximately 3 years.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Arm 1/Magnetic Resonance (MR) Thermal Image Guided Laser Ablation
Number analyzed (Participants) | 15
score on a scale | -2 (0.7)

7. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0)
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: For all participants enrolled over the time frame of the study including follow up time is approximately 65 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1/Magnetic Resonance (MR) Thermal Image Guided Laser Ablation
Number analyzed (Participants) | 15
Participants | 8

ADVERSE EVENTS:
Time Frame: For all participants enrolled over the time frame of the study including follow up time is approximately 65 months.
Arm/Group | Arm 1/Magnetic Resonance (MR) Thermal Image Guided Laser Ablation
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 8/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1/Magnetic Resonance (MR) Thermal Image Guided Laser Ablation (N=15)
Hematuria (Renal and urinary disorders) | 4 (4)
Other, Peyronie's Disease (Reproductive system and breast disorders) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Other, epididymitis (Reproductive system and breast disorders) | 1 (1)
Other, weak stream (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-07-13): https://cdn.clinicaltrials.gov/large-docs/53/NCT01377753/Prot_SAP_000.pdf
  • Informed Consent Form (2015-03-13): https://cdn.clinicaltrials.gov/large-docs/53/NCT01377753/ICF_001.pdf